CLINICAL TRIAL: NCT03673371
Title: Women's-Specific Footwear With Prosthetic Feet
Acronym: WSF
Status: Completed | Type: Observational
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew H. Hansen, Site Principal Investigator, Minneapolis Veterans Affairs Medical Center
Other Study IDs: OP160063
Record Dates: First submitted 2018-08-23; First posted 2018-09-17 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation Above Knee (Injury)
Keywords: Limb Prosthesis; Shoe; Self Concepts
MeSH Terms: conditions — Wounds and Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women Veterans with Lower Limb Amputations: Questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — This is a questionnaire developed by DoD and VA researchers specifically for this study.
  Other Names: "WSF Questionnaire"

SUMMARY:
The purpose of this study is to address footwear challenges unique to women prosthesis users. Comparing the effectiveness of different footwear and prosthesis combinations will help guide clinical decision making regarding the prescription of prosthetic devices, while keeping what the patient wants in mind.

It is expected that these results will be used to generate new knowledge for the development of versatile prosthetic devices that accommodate a user's unique lifestyle while helping the patient to make good progress in rehabilitation.

Investigators will characterize perceived limitations in footwear among women prosthesis users. Investigators think that women prosthesis users will be restricted in footwear choices and clothing choices due to the use of a prosthetic device.

Specifically, investigators expect perceived limitations in footwear will be greater for shoes with higher heels than shoes without heels.

DETAILED DESCRIPTION:
The project involves development, distribution, and analysis of a questionnaire designed to address footwear use among women lower limb prosthesis users. Responses from sixty women with a lower extremity amputation will be targeted. VA participants will be identified by the MVAHCS. These potential participants will receive the IRB-approved survey via mail. Eligible participants include women with unilateral or bilateral lower extremity amputations.

The questionnaire will target the types of footwear worn by prosthesis users and the types of footwear desired to be worn. It will also capture the various types of prosthetic feet worn in each footwear category, amputation type, time spent walking in a prosthetic device, and general satisfaction with the prosthesis function during daily living when worn with shoes.

ELIGIBILITY:
Inclusion Criteria:

* Woman Veteran
* Age 18-80
* Lower Limb Amputation (transtibial, through the knee, transfemoral)
* Eligible to receive care through the VA Health Care System
* Ambulatory and currently using a prosthesis

Exclusion Criteria:

* Syme's Amputation
* Hip Disarticulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women Veterans with Lower Limb Amputation (excluding Syme's and Hip Disarticulation)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Women's-Specific Footwear and Prosthetic Feet Questionnaire | through data collection, an average of one year
  Questionnaire regarding Women Veterans and their use of different types of footwear with prosthetic feet. The subscales are derived from the following scales:Patient Reported Outcome System (PROMIS) Anxiety - 4 Patient Reported Outcome System (PROMIS) Depression - 4 Patient Reported Outcome System - Ability to Participate in Social Roles and Activities Patient Reported Outcome System - Satisfaction with Social Roles and Activities - 4a Amputee Body Image Scale - Revised Prosthetic Limb Users Survey of Mobility Community Participation Index - Importance subscale Community Participation Index - Control subscale Community Participation Index - Frequency index Activities-Specific Balance Confidence Scale Prosthesis Evaluation Questionnaire - Appearance Prosthesis Evaluation Questionnaire - Utility

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Russell Esposito, PhD, Principal Investigator — Extremity Trauma and Amputation Center of Excellence
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized data set will be created and shared under a written agreement that prohibits the recipient from identifying or attempting to re-identify any individual whose data are included in the data set.
Time Frame: Starting 6 months after publication for up to 10 years.
Access Criteria: The Principal Investigator and Site Principal Investigator will review requests for the de-identified final data set. It is possible that the de-identified final data set will be available through PubMed Central.

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Elnitsky CA, Latlief GA, Andrews EE, Adams-Koss LB, Phillips SL. Preferences for rehabilitation services among women with major limb amputations. Rehabil Nurs. 2013 Jan-Feb;38(1):32-6. doi: 10.1002/rnj.62. PMID 23365003
- [Background] Klodd E, Hansen A, Fatone S, Edwards M. Effects of prosthetic foot forefoot flexibility on gait of unilateral transtibial prosthesis users. J Rehabil Res Dev. 2010;47(9):899-910. doi: 10.1682/jrrd.2009.10.0166. PMID 21174254
- [Background] Meier MR, Tucker KA, Hansen AH. Development of inexpensive prosthetic feet for high-heeled shoes using simple shoe insole model. J Rehabil Res Dev. 2014;51(3):439-50. doi: 10.1682/JRRD.2013.01.0010. PMID 25019666